CLINICAL TRIAL: NCT06006845
Title: When to Initiation Antitumor Therapy for Tumor Patients With COVID19 Infection
Brief Title: Time to Initiated Antitumor Therapy for Tumor Patients With COVID19 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wang Bo, Professor, The Seventh Affiliated Hospital of Sun Yat-sen University
Other Study IDs: pan-01
Record Dates: First submitted 2023-08-22; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Tumor; COVID-19
Keywords: Tumor patients; COVID-19; antitumor therapy
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A: Tumor patients infected with COVID-19

SUMMARY:
The goal of this observational study is to study the safety of initiation of antitumor therapy early after nucleic acid test turn negativity in tumor patients infected with COVID-19. The main questions aims to answer are:

* Whether initiation of antitumor therapy early after nucleic acid test turn negativity in tumor patients infected with COVID-19 increases adverse events related to antitumor therapy.
* Whether initiation of antitumor therapy early after nucleic acid test turn negativity in tumor patients infected with COVID-19 increases risk of re-infection of COVID-19.
* How initiation of antitumor therapy early after nucleic acid test turn negativity in tumor patients infected with COVID-19 affects QoL of tumor patients

Participants will be asked to answer the question about:

* the severity and duration of COVID-19 symptoms
* the date of diagnosis of COVID-19
* the date of negative nucleic acid test
* the QoL of life before infection with COVID-19, during infection of COVID-19, after nucleic acid test negativity and receiving antitumor therapy

ELIGIBILITY:
Inclusion Criteria:

* Tumor patients diagnosed with COVID-19 infection at our center from December 1, 2022 to May 31.
* COVID-19 was confirmed by antigen testing or nucleic acid testing.
* Tumor was confirmed by pathology.
* Patients received systemic antitumor therapy after infected with COVID-19.

Exclusion Criteria:

* COVID-19 was not confirmed by antigen testing or nucleic acid testing
* Tumor was not confirmed by pathology
* Patients did not receive systemic antitumor therapy
* Patients died before receiving systemic antitumor therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumor patients infected with COVID-19 from December 1, 2022 to May 31, and received systemic antitumor therapy after infected with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events after antitumor therapy | 28 days after antitumor therapy
  Incidence of adverse events after antitumor therapy, including hematologic toxicity,gastrointestinal adverse event, hepatobiliary adverse events, etc.
Re-infection of COVID-19 | 28 days after antitumor therapy
  Antigen testing or nucleic acid testing positive for COVID-19

SECONDARY OUTCOMES:
Clinical manifestations of COVID-19 in tumor patients | Until nucleic acid testing turn negative
  Symptoms and lab abnormality of COVID-19 in tumor patients

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, Principal Investigator — The Seventh Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong, China